CLINICAL TRIAL: NCT03795428
Title: A Long-Term, Open Label Extension Study of Pemziviptadil (PB1046) Subcutaneous Injections in Pulmonary Arterial Hypertension Subjects Following Completion of Study PB1046-PT-CL-0004
Brief Title: Long-Term, Open Label Extension Study of Pemziviptadil (PB1046) in PAH Subjects Following Completion of Study PB1046-PT-CL-0004
Acronym: VIP Extend
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated: Study drug resupply delayed (Covid-19)
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PB1046-PT-CL-0006
Record Dates: First submitted 2018-12-18; First posted 2019-01-07 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — VIP-ELP fusion molecule PB1046; Injections

STUDY DESIGN:
Intervention Model Description: To protect the blind of the parent study (PB1046-PT-CL-0004), all subjects entering PB1046-PT-CL-0006 will commence dosing at Week 1 on 0.4 mg/kg and will be up-titrated in 0.2 mg/kg increments in an open label fashion for 9 weeks.
Masking Description: Subjects entering the 0006 trial prior to the implementation of this protocol amendment will remain blinded until such time that open label dosing will not unblind the 0004 study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pemziviptadil (PB1046) Injection-OL Active Drug-Up-Titration to Stable Dose (Experimental): Pemziviptadil (PB1046) Injection: Regardless of dose assignment, all subjects will be up-titrated in 0.2 mg/kg weekly increments, beginning with 0.4 mg/kg at Week 1, to the target dose of 1.2 mg/kg or higher depending on safety and tolerability.
  Interventions: Drug: Pemziviptadil (PB1046) Injection

INTERVENTIONS:
Drug: Pemziviptadil (PB1046) Injection — Once-weekly subcutaneous injection

SUMMARY:
This is a multi-center, Phase 2 Long-Term, Open Label Extension (OLE) Study to assess the safety and tolerability of pemziviptadil (PB1046) at an optimally titrated dose. This is a Long-Term, Open label Extension (OLE) Study for subjects with (PAH), having participated in double-blind Study PB1046-PT-CL-0004. The study will include adult subjects previously diagnosed with symptomatic PAH, who are receiving background clinician-directed therapy for PAH.

During this period, subjects will continue to be followed for safety and tolerability, as well as for periodic efficacy, quality of life data and immunogenicity. The study will continue per the schedule of events until such time when pemziviptadil (PB1046) is able to be self-administered, becomes commercially available to the subjects in a particular country or region, or the sponsor terminates the study due to lack of efficacy, safety or other reasons.

DETAILED DESCRIPTION:
Subjects entering this study will enter from the double-blind Study PB1046-PT-CL-0004. The starting dose level of pemziviptadil (PB1046) for all subjects in this parent study was a sub-therapeutic or minimally effective dose (MED) of 0.2 mg/kg, administered by SC injection.

Subjects were randomized into the MED) Group or a dose-titration group. In the dose-titration group, individual subjects were titrated up to their maximum tolerated dose (MTD) in a blinded fashion, with the objective of titrating subjects up to a dose of at least 1.2 mg/kg or higher in the MTD Group, while subjects in the MED Group remained at the MED level of 0.2 mg/kg, and underwent "sham dose-titration" to maintain the blind.

Subjects entering the 0006 trial prior to implementation of this protocol amendment will remain blinded until such time that open label dosing will not unblind the 0004 study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have completed Week 17 / End of Study of PB1046-PT-CL-0004;
* Willing and able to sign a written Informed Consent (IC) prior to all study-related procedures;
* Agrees to use a medically acceptable method of contraception (both male and female patients) throughout the entire study period and continuing for 30 days after their last dose of study drug. if the possibility of conception exists. Medically acceptable methods of contraception include the following: abstinence (not having sex), vasectomy (with confirmed negative sperm counts), condoms and partner using vaginal spermicide and/or cervical cap with spermicide or sponge; oral, implantable, or injectable contraceptives (starting ˃2 months before dosing), diaphragm with vaginal spermicide, intrauterine device, surgical sterilization (˃6 months after surgery). Female subjects ˂45 years of age of non-childbearing potential are defined as being surgically sterile by bilateral tubal ligation, bilateral oophorectomy, or hysterectomy. Female subjects 45to-60 years of age, inclusive, who are post-menopausal for at least 1 year, and have a follicle-stimulating hormone (FSH) level confirmation indicating post-menopausal status, will be considered to be of non-childbearing potential. Female subjects > 60 years of age are considered post-menopausal and of non-childbearing potential;
* Willing and able to understand and follow instructions, return to the study unit for specified study visits; and, be able to participate in the study through the Stable Dose Maintenance Period, at a minimum.

Exclusion Criteria:

* Concomitant medical disorder, condition, or history, that in the opinion of the Investigator, would impair the subject's ability to participate in or complete the requirements of the study;
* Pregnant or lactating female subjects;
* Significant liver dysfunction as measured by any one of the following during participation in PB1046-PT-CL-0004. (If exclusionary laboratory results become available after the subject has enrolled in PB1046-PT-CL-0006 they should be discontinued. a. alanine aminotransferase (ALT) > 3.0 times upper limit of normal (ULN) or; b. aspartate aminotransferase (AST) > 3.0 times ULN or; c. serum bilirubin ≥ 1.6 mg/dL.
* Recent history of substance abuse that, in the opinion of the Investigator, would impair the subject's ability to participate in or complete the requirements of the study;
* In the opinion of the principal investigator (PI), any major surgical procedure within 90 days, or a planned surgical procedure during the study period; which would impact participation in PB1046-PT-CL-0006.
* Other new medical or psychiatric conditions which, in the opinion of the Investigator, would place the subject at increased risk, would preclude obtaining voluntary consent, or would confound the objectives of the study;
* Known hypersensitivity to study drug or any of the excipients of the drug formulation.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
Incidence of Clinical Laboratory Abnormalities | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
Change in Diastolic Blood Pressure from baseline | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
Change in Systolic Blood Pressure from baseline | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
Change in Oral Body Temperature from baseline | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
Change in Respiratory Rate from baseline | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
Change in Heart Rate from baseline | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
12-Lead ECG - Incidence of clinically significant abnormal ECG findings as measured by 12 Lead ECG | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
Incidence of Immunogenicity | Duration of extension study - Starting up to 30 days prior to first dose of study drug in original study (PB1046-PT-CL-0004/0005) and completing 28 days after last dose.
  Incidence of positive immunogenicity results after receipt of study drug

SECONDARY OUTCOMES:
Survival | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
Change from baseline in 6MWD (6 minute walk distance test) | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
  Measured in meters walked in 6 minutes.
Change from baseline in NT-proBNP | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
Change from baseline in NYHA/WHO Functional Class (FC) | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
Change from baseline in emPHasis-10 (Health Related Quality of Life) score | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
  Scores, which assess breathlessness, fatigue, control and confidence, range from 0 to 50, higher scores indicate worse quality of life.
Change from baseline in Borg Dyspnea Index (BDI) | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
  BDI scale as measured from 0 to 10 (0 being no breathlessness and 10 being maximal breathlessness)
Incidence of Clinical Worsening | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
  As defined by any one of the following: 1. All cause mortality; 2. Hospitalization due to worsening PAH; 3. Initiation of parenteral prostacyclin; 4. Any three of the following: 15% decrease in 6MWD, Functional class III or IV symptoms, Addition of PAH therapy, Worsening right heart failure
Change in REVEAL Registry Risk Calculator Score | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
  Risk scores range from 0 (Lowest risk) to 22 (Highest risk) in PAH subjects

OTHER OUTCOMES:
Change in pulmonary artery pressure from baseline | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
  PB1046-PT-CL-0005 subjects only as measured by CardioMEMS device
Change in cardiac index from baseline | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
  PB1046-PT-CL-0005 subjects only as measured by CardioMEMS device
Change in total pulmonary resistance from baseline | Duration of extension study - Starting the day of first dose and completing 28 days after last dose.
  PB1046-PT-CL-0005 subjects only as measured by CardioMEMS device

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of California San Diego, La Jolla, California
  - University of California - Davis, Sacramento, California
  - University of Miami - Pulmonary Research Center, Miami, Florida
  - Emory University, The Emory Clinic, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No